CLINICAL TRIAL: NCT04441021
Title: Feasibility Assessment of Risk Stratification and Oral Challenge in Hospitalized Children at Low Risk for Antibiotic Allergy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, James Antoon, Assistant Professor, Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 200251-2; 5K12HL137943-03 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Penicillin Allergy Risk Stratification and Evaluation: This standard of care intervention will provide an antibiotic allergy risk stratification assessment and subsequent amoxicillin oral challenge in patients who stratify as low risk for true allergy
  Interventions: Other: Penicillin Allergy Risk Stratification and Evaluation

INTERVENTIONS:
Other: Penicillin Allergy Risk Stratification and Evaluation — This standard of care intervention will provide an antibiotic allergy risk stratification assessment and subsequent amoxicillin oral challenge in patients who stratify as low risk for true allergy

SUMMARY:
Children are often reported to have antibiotics allergies, with approximately 10% of the US population labeled as allergic to an antibiotic. Recent studies have demonstrated that a large majority of children with a penicillin allergy label do not have a true IgE-mediated allergy. Appropriately delabeling antibiotic allergies has been shown to improve patient care outcomes and lower health care costs. However, efforts to implement these assessments in practice are lacking, particularly in the hospital setting. Therefore, there is a need for hospital-based risk assessment and delabeling strategies for hospitalized children. The investigator's objective is to determine the feasibility of implementing a hospital-based approach to penicillin allergy risk stratification and evaluation of patients at low-risk for true allergy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Vanderbilt children's hospital admitted to a Pediatric Hospital Medicine service with a penicillin allergy reported in their chart who are medically stable

Exclusion Criteria:

* Known pregnancy
* Patients without a primary care provider

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals admitted to Vanderbilt children's hospital admitted to a Pediatric Hospital Medicine service with a penicillin allergy reported in their chart who are medically stable
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | Within 2 weeks of hospital discharge
  Qualitative survey to assess feasibility of intervention

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | Within 2 weeks of hospital discharge
  Qualitative survey to assess acceptability of intervention
Intervention Appropriateness Measure | Within 2 weeks of hospital discharge
  Qualitative survey to assess appropriateness of intervention

CONTACTS AND LOCATIONS:
Overall Officials: James Antoon, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antoon JW, Grijalva CG, Grisso AG, Stone CA, Johnson J, Stassun J, Norton AE, Kripalani S, Williams DJ. Feasibility of a Centralized, Pharmacy-Led Penicillin Allergy Delabeling Program. Hosp Pediatr. 2022 Jul 1;12(7):e230-e237. doi: 10.1542/hpeds.2021-006369. PMID 35678128